CLINICAL TRIAL: NCT00039936
Title: Treatment of Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMitchell (completed)
Record Dates: First submitted 2002-06-17; First posted 2002-06-19 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Bulimia; Obesity
Keywords: Binge Eating; Obesity; Cognitive; Behavior
MeSH Terms: conditions — Bulimia; Obesity; Behavior

INTERVENTIONS:
Behavioral: Cognitive Behavior Treatment
Behavioral: Self Help
Behavioral: Partial Self Help

SUMMARY:
This is a multicenter (2 sites) randomized trial evaluating three group treatment models for subjects with binge eating disorder. One model is a cognitive behavior treatment (CBT) group, one is partial self help, and one is self help only.

ELIGIBILITY:
* Meet binge eating disorder (BED) Criteria
* Not psychotic
* Not in other treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2002-02

CONTACTS AND LOCATIONS:
Locations (1):
- NRI, Fargo, North Dakota, United States

REFERENCES:
- See also: Host Institution — http://www.nrifargo.com